CLINICAL TRIAL: NCT02426541
Title: An 8-week, Single Centre, Randomized, Parallel-group, Double-blind, Placebo Controlled Phase IV Study to Evaluate Dapagliflozin 10 mg Once Daily Effects on Insulin Resistance in Subjects With Type 2 Diabetes Mellitus
Brief Title: Effects of Dapagliflozin 10 mg on Insulin Resistance in Patients With Type 2 Diabetes Mellitus
Acronym: DERISC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Antaros Medical (Industry); Bioventure Hub (Unknown); 43183 Mölndal (Unknown); Sweden (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D1690C00025; 2014-005377-36 (EudraCT Number)
Record Dates: First submitted 2015-04-22; First posted 2015-04-27 (Estimated); Results first posted 2018-02-05 (Actual); Last update posted 2018-02-05 (Actual); Status verified 2017-07

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes Mellitus; Dapagliflozin; Placebo; Insulin resistance; Insulin sensitivity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Insulin Resistance | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dapagliflozin (Experimental): Dapagliflozin Once Daily 10 mg
  Interventions: Drug: Dapagliflozin
- Placebo (Placebo Comparator): Matching placebo for Dapagliflozin Once Daily 10 mg
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin — Dapagliflozin 10 mg Tablets, Oral, Once Daily, 8 weeks
  Other Names: Forxiga, Farxiga
  Arms: Dapagliflozin
Drug: Placebo — Matching placebo to Dapagliflozin 10 mg Tablets, Oral, Once Daily, 8 weeks
  Arms: Placebo

SUMMARY:
This is an 8-week, single centre, randomized, parallel-group, double-blind, placebo-controlled Phase IV study to evaluate the effect of dapagliflozin on tissue specific insulin sensitivity in patients with Type 2 diabetes mellitus

ELIGIBILITY:
Main Inclusion Criteria:

1. Provision of signed informed consent prior to any study specific procedures.
2. Female or male aged 35 to 70 years inclusive with suitable veins for cannulation or repeated venipuncture
3. Type 2 Diabetes mellitus defined as HbA1c of ≥ 6.5% and ≤ 10.5%.
4. Stable (≥ 3 months) T2D treatment with metformin and/or metformin+dipeptidyl peptidase-4 inhibitors (DPP-IV)
5. Body mass index (BMI) ≤ 40 kg/m2.
6. Female subjects must be of non-childbearing potential, meeting at least one of the following criteria:

   1. Hysterectomized females
   2. Postmenopausal women, defined as women who have not had a menstrual period within 1 year

Main Exclusion Criteria:

1. Any condition that is contraindicated with MRI such as, but not limited to, having a pacemaker or claustrophobia.
2. Volume depleted patients. Patients at risk for volume depletion due to co-existing conditions or concomitant medications, such as loop diuretics should have careful monitoring of their volume status.
3. Recent Cardiovascular Events in a patient:

   * Acute Coronary Syndrome (ACS) within 2 months prior to enrolment
   * Hospitalization for unstable angina or acute myocardial infarction within 2 months prior to enrolment
   * Acute Stroke or Transient Ischemic Attack (TIA) within two months prior to enrolment
   * Less than two months post coronary artery revascularization
4. Congestive heart failure defined as New York Heart Association (NYHA) class IV, unstable or acute congestive heart failure.
5. Blood pressure at enrolment: Systolic BP ≥165 mm Hg and/or diastolic BP ≥100 mm Hg
6. Any clinically significant illness, medical or surgical procedure or trauma within 4 weeks of the first administration of the investigational product.
7. On insulin, GLP-1 or other oral antidiabetic drug treatment (metformin or both metformin and DPP-IV allowed) or using other medications known to affect glucose metabolism.
8. Any clinically significant abnormalities in physical examination, Electrocardiography (ECG) or clinical chemistry results as judged by the investigator. The following specific exclusion criteria apply to the selected Clinical Chemistry results:

   1. Creatinine clearance <60mL/min (estimated with Cockroft-Gault formula).
   2. Severe hepatic insufficiency and/or significant abnormal liver function defined as aspartate aminotransferase (AST) >3x upper limit of normal (ULN) and/or alanine aminotransferase (ALT) >3x ULN.
   3. Total bilirubin (TB) >2.0 mg/dL (34.2 µmol/L).
9. Body weight loss greater than 5% within 3 months prior to Visit 1.
10. Previous PET scan
11. History of or presence of (as found at Visit 1) any clinically significant disease, disorder or condition which, in the opinion of the investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study.

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2015-03-23 (Actual); Primary Completion 2016-04-28 (Actual); Study Completion 2016-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pirjo Nuutila, MD, PhD, Professor, Principal Investigator — Turku PET Centre, Turku, Finland
Locations (1):
- Research Site, Turku, Finland

REFERENCES:
- [Derived] Latva-Rasku A, Honka MJ, Kullberg J, Mononen N, Lehtimaki T, Saltevo J, Kirjavainen AK, Saunavaara V, Iozzo P, Johansson L, Oscarsson J, Hannukainen JC, Nuutila P. The SGLT2 Inhibitor Dapagliflozin Reduces Liver Fat but Does Not Affect Tissue Insulin Sensitivity: A Randomized, Double-Blind, Placebo-Controlled Study With 8-Week Treatment in Type 2 Diabetes Patients. Diabetes Care. 2019 May;42(5):931-937. doi: 10.2337/dc18-1569. Epub 2019 Mar 18. PMID 30885955

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 55 subjects were enrolled and 32 subjects were randomised and treated. One participant was withdrawn prior to study completion. Thirty-one participants completed the study and attended all visits.
Groups:
- Dapagliflozin 10 MG: Dapagliflozin 10 MG added to stable metformin, dipeptidyl pepdidase-4 (DPP-IV) inhibitor, or sulphonylurea alone or in combination with either metformin or DPP-IV inhibitor antidiabetic medication.
- Placebo: Placebo added to stable metformin, dipeptidyl pepdidase-4 (DPP-IV) inhibitor, or sulphonylurea alone or in combination with either metformin or DPP-IV inhibitor antidiabetic medication.
Period: Overall Study
Arm/Group | Dapagliflozin 10 MG | Placebo
Started | 16 | 16
Completed | 15 | 16
Not Completed | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Population: Population represents the full analysis set which includes all randomised subjects who received at least one dose of study with a non-missing baseline value and at least one post-baseline value for at least one primary or secondary efficacy variable during the double-blind period.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dapagliflozin 10 MG | Placebo | Total
Number analyzed (Participants) | 15 | 16 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] — Age of participant
  years | 62.1 (8.4) | 59.9 (7.4) | 61.0 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 13 | 12 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 15 | 16 | 31
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Secondary Outcome: Adjusted Change in Adipose Tissue Insulin-stimulated Glucose Uptake
Description: Change in adipose tissue insulin-stimulated glucose uptake assessed by hyperglycemic-euglycemic clamp using F-FDG PET
Time Frame: Baseline to Week 8
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: umol/min/kg
Arm/Group | Dapagliflozin 10 MG | Placebo
Number analyzed (Participants) | 15 | 16
umol/min/kg | 1.04 (1.50) | -0.64 (1.36)
Statistical Analysis 1: Comparison: Dapagliflozin 10 MG vs Placebo; Test type: Superiority or Other; p = 0.3794, ANCOVA; Adjusted for sex and baseline; Mean Difference (Final Values) = 1.68, 95% CI 2-sided [-2.18 to 5.54]

2. Secondary Outcome: Adjusted Change in Liver Insulin-stimulated Glucose Uptake From Baseline to Week 8
Description: Adjusted change in liver insulin-stimulated glucose uptake assessed by hyperglycemic-euglycemic clamp using F-FDG PET
Time Frame: Baseline to Week 8
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: umol/min/kg
Arm/Group | Dapagliflozin 10 MG | Placebo
Number analyzed (Participants) | 15 | 16
umol/min/kg | 0.27 (1.74) | 1.59 (1.52)
Statistical Analysis 1: Comparison: Dapagliflozin 10 MG vs Placebo; Test type: Superiority or Other; p = 0.5317, ANCOVA; Adjusted for sex and baseline; Mean Difference (Final Values) = -1.32, 95% CI 2-sided [-5.60 to 2.96]

3. Primary Outcome: Adjusted Change From Baseline in Skeletal Muscle Insulin-stimulated Gluocose Uptake
Description: Adjusted change from baseline in skeletal muscle insulin-stimulated gluocose uptake (umol/min/kg)
Time Frame: From baseline to Week 8
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: umol/min/kg
Arm/Group | Dapagliflozin 10 MG | Placebo
Number analyzed (Participants) | 15 | 16
umol/min/kg | 0.28 (1.23) | 0.28 (1.13)
Statistical Analysis 1: Comparison: Dapagliflozin 10 MG vs Placebo; Test type: Superiority or Other; p = 0.9984, ANCOVA; Adjusted for sex and baseline; Mean Difference (Final Values) = -0.0030, 95% CI 2-sided [-3.07 to 3.07]

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Dapagliflozin 10 MG | Placebo
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 6/16 | 7/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dapagliflozin 10 MG (N=16) | Placebo (N=16)
Balanitis candida (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Astenia (General disorders) | 0 (0) | 1 (1)
Thirst (General disorders) | 1 (1) | 0 (0)
Blood glucose decreased (Investigations) | 1 (1) | 0 (0)
Polyuria (Renal and urinary disorders) | 4 (4) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All drafts of proposed publications, written reports, training materials, advertisements and similar documents related to the Services and intended to be communicated or published to any third party ("Communications") must be submitted to Antaros for AstraZeneca's review and approval prior to dissemination.